CLINICAL TRIAL: NCT00394472
Title: A Randomized, Double-blind, Placebo Controlled, Phase IIA Study to Assess the Effect on Gastroesophageal Reflux Disease (GERD) Symptoms, Pharmacokinetics, Safety and Tolerability of 4 Weeks Treatment With AZD3355 65 mg Bid as add-on Treatment to a Proton Pump Inhibitor (PPI) in Patients With an Incomplete Response to PPI.
Brief Title: Symptom Improvements in Gastroesophageal Reflux Disease (GERD) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D9120C00011; EUDRACT No 2006-003541-16
Record Dates: First submitted 2006-10-31; First posted 2006-11-01 (Estimated); Results first posted 2013-03-18 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-02

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: Heartburn; Patient reported symptoms; Proton pump inhibitor
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn | interventions — lesogaberan

INTERVENTIONS:
Drug: AZD3355
  Other Names: Lesogaberan

SUMMARY:
The purpose of this study is to estimate the effect of AZD3355 as an add-on treatment to a Proton Pump Inhibitor (PPI) on Gastroesophageal reflux disease (GERD) symptoms in patients with an incomplete response to PPI treatment.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* At least 6 months history of Gastroesophageal reflux disease (GERD) symptoms
* Continuous treatment with Proton Pump Inhibitor (PPI)
* Ability to read and write

Exclusion Criteria:

* Prior surgery of the upper gastrointestinal (GI) tract
* History of clinically significant diseases other than GERD
* Need for concomitant medication with drugs that may influence gastrointestinal symptoms

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2006-11; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Göran Hasselgren, MD, Study Director — AstraZeneca; Guy Boeckxstaens, MD, Principal Investigator — Academisch Medisch Centrum Universiteit van Amsterdam
Locations (38):
- Research Site, Adelaide, Australia
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Eupen
  - Research Site, Wilrijk
- France (5):
  - Research Site, Alès
  - Research Site, Angers
  - Research Site, Bordeaux
  - Research Site, Lyon
  - Research Site, Nantes
- Germany (8):
  - Research Site, Cologne
  - Research Site, Koblenz
  - Research Site, Ludwigshafen
  - Research Site, München
  - Research Site, Oelde
  - Research Site, Potsdam
  - Research Site, Wangen
  - Research Site, Wiesbaden
- Hungary (8):
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Nagykanizsa
  - Research Site, Pécs
  - Research Site, Siófok
  - Research Site, Szeged
  - Research Site, Szombathely
  - Research Site, Vác
- Research Site, Amsterdam, Netherlands
- Norway (8):
  - Research Site, Ålesund
  - Research Site, Bergen
  - Research Site, Levanger
  - Research Site, Oslo
  - Research Site, Rud
  - Research Site, Stavanger
  - Research Site, Tromsø
  - Research Site, Trondheim
- Romania (4):
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Satu Mare
  - Research Site, Târgu Mureş

REFERENCES:
- [Derived] Boeckxstaens GE, Beaumont H, Hatlebakk JG, Silberg DG, Bjorck K, Karlsson M, Denison H. A novel reflux inhibitor lesogaberan (AZD3355) as add-on treatment in patients with GORD with persistent reflux symptoms despite proton pump inhibitor therapy: a randomised placebo-controlled trial. Gut. 2011 Sep;60(9):1182-8. doi: 10.1136/gut.2010.235630. Epub 2011 Mar 14. PMID 21402616

RESULTS

PARTICIPANT FLOW:
Groups:
- AZD3355: AZD3355 capsules 65 mg bid
- Placebo: Placebo capsules bid
Period: Overall Study
Arm/Group | AZD3355 | Placebo
Started | 122 | 122
Completed | 113 | 111
Not Completed | 9 | 11
Not completed — Protocol Violation | 1 | 3
Not completed — incorrect enrolment | 4 | 2
Not completed — Adverse Event | 4 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD3355 | Placebo | Total
Number analyzed (Participants) | 122 | 122 | 244
Age Continuous [Mean (Standard Deviation); unit: years] | 51.1 (11.9) | 48.7 (12.6) | 49.9 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 31 | 82
  Male | 71 | 91 | 162

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Most One Day With Not More Than Mild Intensity of the Symptoms 'a Burning Feeling Behind the Breastbone' and 'Unpleasant Movement of Material Upwards From the Stomach' During the Last Seven Days of Treatment
Description: Symptom intensity rated by participants twice daily on a six-graded Likert scale (Did not have; Very mild; Mild; Moderate; Moderately severe; Severe) using an electronic Reflux Disease Questionnaire (RDQ) diary
Time Frame: Twice daily during the last seven days on treatment
Measure: Number; unit: Participants
Arm/Group | AZD3355 | Placebo
Number analyzed (Participants) | 114 | 118
Participants | 17 | 8

2. Secondary Outcome: Plasma Concentration (µmol/L) of AZD3355 Analysed From Blood Sample Taken in the Interval One to Two Hours After the First Intake of AZD3355 65 mg Capsule
Time Frame: An interval of one to two hours after the first intake of AZD3355 65 mg capsule
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | AZD3355 | Placebo
Number analyzed (Participants) | 122 | 0
μmol/L | 0.96 (0.74) |

ADVERSE EVENTS:
Arm/Group | AZD3355 | Placebo
Serious Adverse Events (participants affected / at risk) | 2 | 0
Other Adverse Events (participants affected / at risk) | 28 | 19
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | AZD3355 | Placebo
Hypertension (Vascular disorders) | 1/122 | 0/122
Appendicitis (Infections and infestations) | 1/122 | 0/122
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | AZD3355 | Placebo
DIARRHOEA (Gastrointestinal disorders) | 13/122 | 4/122
NAUSEA (Gastrointestinal disorders) | 9/122 | 4/122
FATIGUE (General disorders) | 7/122 | 7/122
PARAESTHESIA (Nervous system disorders) | 10/122 | 6/122

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AZ shall have 30 days from the proposed final manuscript for any disclosure to review it and may within such time require that submission for publication/disclosure be delayed in order for AZ to file patent applications. If study site/investigator requests permission to publish data(incl oral presentations) it is to be agreed with AZ before publ.